CLINICAL TRIAL: NCT03432910
Title: Study of Application of Forced Breath Technique While CPAP Therapy for Apnea Classification
Brief Title: Application of Forced Breath Technique While CPAP Therapy for Apnea Classification
Acronym: FBT-CPAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heinen und Löwenstein GmbH & Co. KG (Industry)
Collaborators: Löwenstein Medical Technology (Unknown)
Responsible Party: Sponsor
Organization: Heinen (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-pLINE-FBT-C
Record Dates: First submitted 2018-02-05; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Sleep Apnea, Obstructive; Sleep Apnea, Central
Keywords: Forced Breath Technique; auto-CPAP; CPAP; Obstructive sleep apnea; central sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea, Central

STUDY DESIGN:
Intervention Model Description: Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Other): Participants of the study undergo the standard stages of the clinical routine within a PAP therapy setting: a diagnostic night followed by one or two treatment nights.
  Interventions: Other: CPAP Titration using a Bilevel S/T mode with minimal pressure support and background rate

INTERVENTIONS:
Other: CPAP Titration using a Bilevel S/T mode with minimal pressure support and background rate — The study performs within clinical routine with this exception that instead of the usually applied CPAP mode a modified BiLevel S/T mode is used. The modified BiLevel S/T mode meets the same requirements as the CPAP mode while providing the Forced Breath Technique to classify apneas as central or obstructive.

SUMMARY:
This study analyzes the application of the Forced Breath Technique (FBT) to classify apneas during CPAP therapy with a prismaLAB (device name) therapy device.

In this study the BiLevel ST (Spontaneous / Timed) therapy mode of the prismaLAB device is reduced to a CPAP pressure profile with exhalation relief by minimization of the pressure gap between exhalation and inhalation pressure.

The FBT based apnea classification of the devices firmware is matched with the by hand scoring of the polysomnographic data that is usually used to evaluate the quality of patients sleep.

DETAILED DESCRIPTION:
Obstructive sleep-disordered breathing is usually treated by positive airway pressure (PAP) therapy with respective devices.The devices detect, classify and store respiratory events as apneas, hypopneas and snoring to adapt the therapy pressure according to patients needs and/ or to validate therapy efficacy.

Since several years the Forced Breath Technique (FBT) is standard practice in PAP devices with a BiLevel pressure profile and a background rate to classify apneas as central or obstructive. In case of an interruption of the respiratory flow within an apnea the devices background rate applies so called "mandatory breaths" with neither a manually or by device defined pressure gap between exhalation and inhalation pressure (PDIFF). If a mandatory breath generates respiratory flow patients airways are open and the patient gets ventilated. In this case the detected apnea is classified as central. If a mandatory breath generates no or insufficient respiratory flow patients airways are impassable and the apnea is classified as an obstructive event.

Usually the size of the applied therapeutic pressure gap PDIFF is >= 4 hPa. If patients airways are open the mandatory breaths with PDIFF>= 4 hPa generate an obvious flow that submits a valid classification of apneas. Therefore the pressure gap should be preferably large. So, too, the pressure gap size should be defined as small as possible to prevent the impairment of patients sleep quality.

This pilot study targets to analyze if the application of FBT with a minor gap between inhalation and exhalation pressure (IPAP [inspiratory positive airway pressure] - EPAP [expiratory positive airway pressure] = PDIFF = 1,0 to 2,0 hPa) qualifies for an equal classification of apneas as with a PDIFF >= 4 hPa. Subsequently it serves to define the minimum size of this pressure gap.

To this effect the study is subdivided in to phases: an optimization phase and an evaluation phase.

The optimization phase targets to define the PDIFF size that enables the valid classification of apneas. The evaluation phase serves to compute the accuracy of the classification, the optimized algorithm and the determined classification criteria. Therefore this phase only takes place if the optimization phase yielded a result.

The optimization phase starts with a PDIFF of 1,5 hPa. If this PDIFF serves the purpose, the phase continues with a PDIFF of 1,0 hPa to analyze if a smaller pressure gap yields similar results. Otherwise the phase continues with a PDIFF of 2,0 hPa. Afterwards the optimization phase ends.

The review of the matching of the apneas classified by the device vs the manual scoring takes place after the synchronization of both sources.

Within every PDIFF round in the optimization phase patient recruitment takes place as long as at least 60 obstructive and 60 central apneas have been collected. To guarantee an equal dispersion of apneas on the patient population only 10 obstructive and 10 central apneas of each patient go down in the pool of apneas of the respective PDIFF round. The apnea extraction is made by randomization.

The evaluation phase runs with the determined PDIFF until at least 80 obstructive and 80 central apneas are collected.

The data evaluation occurs by use of descriptive statistics and based on fourfold tables.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of sleep-disordered breathing (AHI >= 15/h)
* ensued or indicated CPAP titration within a routine PAP therapy setting
* age >= 18 years
* presence of written informed consent
* in case of therapy control or repeated participation: total number of apneas in the ensued treatment night was > 10

Exclusion Criteria:

* written informed consent is missing
* Participation in another clinical trial that influences the initiation of (auto) CPAP treatment by specifications of device settings or titration procedure
* NYHA (New York Heart Association) class III or IV
* acute cardiac decompensation
* severe arrhythmia
* severe hypotension, particularly in combination with intravascular volume depletion
* severe epistaxis
* high risk of barotrauma
* decompensated pulmonary conditions
* pneumothorax or pneumomediastinum
* pneumocephalus
* cranial trauma
* status following brain surgery or surgical intervention on the pituitary gland or the middle/inner ear
* acute sinus infection (sinusitis), middle ear infection (otitis media) or perforated eardrum
* dehydration

Exclusion Criteria Statistical Evaluation:

Data of patients who completed the study protocol will be excluded from statistical analysis if one of the following criteria applies:

* there is leakage of > 50 l/min for
* application of incorrect device settings
* insufficient data quality of PSG (Polysomnography) -acquisition
* the device was applied outside range of indication
* data of diagnostic night are not acquired as a PSG
* informed consent isn´t present
* the total number of apneas during the treatment night with BiLevel ST is < 10

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-03-24 (Actual); Primary Completion 2018-02-23 (Estimated); Study Completion 2018-03-29 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the mapping of apneas based on the Forced Breath Technique compared to the manual scoring of polysomnographic data | 1 night (= first treatment night)

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nilius, PD Dr. med., Principal Investigator — HELIOS Klinik Hagen Ambrock
Locations (1):
- HELIOS Klinik, Hagen, North Rhine-Westphalia, Germany